CLINICAL TRIAL: NCT06137300
Title: Safety and Efficacy of Urinary Kallidinogenase for Large Artery Atherosclerosis Acute Ischemic Stroke：a Multicentre, Prospective, Randomised, Open-label, Blinded-Endpoint Trial
Brief Title: Safety and Efficacy of Urinary Kallidinogenase for Large Artery Atherosclerosis Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of the First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TK-LAA
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke, Urinary Kallidinogenase
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinary Kallidinogenase group (Experimental): Patients are treated with urinary kallidinogenase and guideline-prescribed basic medical therapy.
  Interventions: Drug: Urinary kallidinogenase for injection
- Control group (Other): Patients are only treated with guideline-prescribed basic medical therapy.
  Interventions: Other: Guideline-prescribed medical therapy

INTERVENTIONS:
Drug: Urinary kallidinogenase for injection — Urinary kallidinogenase 0.15PNA once daily for 7 days.
  Other Names: Guideline-prescribed medical therapy
  Arms: Urinary Kallidinogenase group
Other: Guideline-prescribed medical therapy — Guideline-prescribed medical therapy
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of urinary kallidinogenase treatment in patients with large artery atherosclerotic acute ischemic stroke.

DETAILED DESCRIPTION:
Currently, evidence regarding the safety and efficacy of urinary kallidinogenase treatment in patients with acute ischemic stroke lacks, and few of related studies were large-scale and high-quality. Thus, this study was designed to evaluate the safety and efficacy of urinary kallidinogenase treatment in patients with large artery atherosclerotic acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Acute anterior circulation large artery atherosclerotic cerebral infarction (according to TOAST classification) within 48h of onset; NIHSS score ≥6, ≤15;
3. Moderate to severe stenosis or occlusion of offending vessels;
4. The mRS Score ≤2 before onset;
5. Subjects or their legal representatives agreed to the treatment and signed the informed consent form.

Exclusion Criteria:

1. Transient ischemic attack;
2. Patients who planned or had received emergency reperfusion therapy (including intravenous thrombolysis and emergency thrombectomy);
3. Severe disturbance of consciousness:GCS ≤8;
4. Patients who previously received angiotensin-converting enzyme inhibitor (ACEI) drugs regularly;
5. Refractory hypertension: systolic blood pressure ≥200 mmHg or diastolic blood pressure ≥110 mmHg; hypotension: systolic blood pressure < 90 mmHg or diastolic blood pressure < 60 mmHg;
6. Liver dysfunction (ALT/AST >1.5 × upper limit of normal [ULN]), renal dysfunction (Cr >1 × ULN);
7. Coagulopathy (prolonged INR (>1.5) or prolonged APTT (>2 folds);
8. Cardioembolic stroke or high-risk factors of cardioembolic stroke identified by investigators (atrial fibrillation, cardiac mural thrombus, cardiomyopathy, etc.);
9. Special populations such as pregnant and lactating women, patients with life expectancy less than 3 months, or patients unable to complete the study for other reasons;
10. Unwilling to be followed up or poor treatment compliance;
11. Participating in other clinical investigators, or had participated in other clinical investigators within 3 months before enrollment;
12. Other conditions considered by the investigator to be inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-2 at 90 days | 90 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) at 7days. | 7days
  National Institute of Health stroke Scale (NIHSS) ranged from 0 to 42, a low value represents a better outcome.
Incidence of ischemic stroke within 90 days. | 0-90days
  Including recurrent and new ischemic stroke.
Adverse events occurring in the course of the treatment. | 0-7days
  Including all adverse events, severe adverse events and urinary kallidinogenase related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD,PhD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China